CLINICAL TRIAL: NCT01081106
Title: Low Level Laser Therapy for Hair Preservation With Chemotherapy for Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 09CC2; STU00021813 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-02-19; First posted 2010-03-05 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-Level Laser Therapy (Other)
  Interventions: Procedure: Low-Level Laser Therapy

INTERVENTIONS:
Procedure: Low-Level Laser Therapy — A LLLT device at 670 nm will be used for light application using lasers affixed in a rotating helmet apparatus. Treatment will be given twice weekly prior to commencing chemotherapy and will be administered once a week until one week after the last chemotherapy.
  administration.

SUMMARY:
The purpose of this study is to see whether low level laser therapy can help maintain normal hair growth on the scalp in people receiving chemotherapy, which is generally associated with hair loss.

DETAILED DESCRIPTION:
Chemotherapy is a common treatment given to patients with breast cancer. Many chemotherapy drugs cause rapid hair loss. While hair loss is temporary, this side effect is a significant concern for patients. Low level laser therapy has been shown to help make hair grow. It is hoped that it may stop hair loss from occurring.

Participants will be receiving 20 to 30 minute laser sessions to their scalp twice a week beginning two weeks before treatment begins until one week past the last chemotherapy session. . Photographs will be taken during each study participant's initial visit, during treatment visits, and one month following the final chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have breast cancer and must be starting chemotherapy with Adriamycin or a taxane-based therapy.
* Participants must be 18 years old or older
* Participants must be female
* Participant must agree to comply with therapeutic and follow-up schedule.
* Patient must signed informed consent form.

Exclusion Criteria:

* Participants cannot have sensitivity to the laser light.
* Participants cannot have used any topical or oral products to grow hair within 3 months of enrollment to this study.
* Participants cannot be pregnant, lactating or planning on pregnancy during therapeutic schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
10 Point Scale to evaluate hair loss | Photographs evaluated weekly during treatment, one month post chemotherapy
  The primary objective is to evaluate the ability of Low-Level Laser Therapy (LLLT) to prevent chemotherapy induced alopecia in women receiving adjuvant chemotherapy for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Van Roenn, MD, Principal Investigator — Northwestern University